CLINICAL TRIAL: NCT04569617
Title: Autonomic Modulation Recovery After Acute Resistance Exercise in Different Intensities and Body Segments
Brief Title: Autonomic Modulation Recovery After Acute Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 34303014.6.0000.5515
Record Dates: First submitted 2020-08-28; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Resistance Training
Keywords: resistance training; autonomic modulation; heart rate; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a cross-over clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- upper limb endurance protocol (Active Comparator): UL endurance protocol - elbow flexion
  Interventions: Other: Resistance Training - UL endurance protocol
- upper limb strength protocol (Active Comparator): UL strength protocol - elbow flexion
  Interventions: Other: Resistance Training - UL strength protocol
- lower limb endurance protocol (Active Comparator): LL endurance protocol - knee extension
  Interventions: Other: Resistance Training - LL endurance protocol
- lower limb strength protocol (Active Comparator): LL strength protocol - knee extension
  Interventions: Other: Resistance Training - LL strength protocol

INTERVENTIONS:
Other: Resistance Training - UL endurance protocol — UL endurance protocol - 2 series of 20 repetitions, elbow flexion at 40% of the maximum test force of 1 maximum repetition, (recovery 1 minutes between sets).
  Arms: upper limb endurance protocol
Other: Resistance Training - UL strength protocol — UL strength protocol - 2 series of 8 repetitions, elbow flexion at 80% of the maximum test force of 1 maximum repetition, (recovery 1 minutes between sets).
  Arms: upper limb strength protocol
Other: Resistance Training - LL endurance protocol — LL endurance protocol - 2 series of 20 repetitions, elbow flexion at 40% of the maximum test strength of 1 maximum repetition, (recovery 1 minutes between sets).
  Arms: lower limb endurance protocol
Other: Resistance Training - LL strength protocol — LL strength protocol - 2 series of 8 repetitions, knee extension at 80% of the maximum test force of 1 maximum repetition, (recovery 1 minutes between sets).
  Arms: lower limb strength protocol

SUMMARY:
To analyze the autonomic behavior in recovery post-acute resistance exercise performed in different intensities and body segments.

DETAILED DESCRIPTION:
Resistance training (RT) is recommended to people with different health condition. RT is recognized as safe and effective method of increasing muscle strength, physical fitness, muscle mass, and overall cardiovascular health. The magnitude of the RT effects is associated with the structure of the training program. Understanding these aspects may provide guidance for the RT prescription while reducing potential risk of cardiovascular events associated with the recovery period after exercise. The objective of the study is to compare the acute responses of the Autonomic Nervous System post RT performed with different intensities (endurance and strength) in different body segments (UL and LL). Our hypothesis is that different intensities and body segments influence the acute responses of the ANS in the post RT recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Graduate students,
* Age between 18 to 30 years
* Healthy men, the Physical Activity Readiness Questionnaire (PAR-Q) was used to determine safety and possible risk of exercising based on participants' health history, the according American College of Sports Medicine, 2010.
* Trained men, the International Physical Activity Questionnaire (IPAQ) was used to determine participants' physical activity level.

Exclusion Criteria: Participants who did not attend all the RT protocols and those with HR record with error higher than 5% (ectopic beats) will be excluded.

-

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2015-01-20 (Actual)

PRIMARY OUTCOMES:
Acute responses of the Autonomic Nervous System post Resistance Training of the time-domain indices of Heart Rate Variability | the moments before and immediately after Resistance Training, performed with different intensities (endurance and strength) and body segments (UL and LL).
  Understand the effect of acute responses of the time-domain indices of Heart Rate Variability, RMSSD, and SDNN, comparing the behavior of these indices of in rest periods and immediate recovery after effort. Besides, to analyze the changes observed when applying different training intensities (endurance protocol 40% 1RM, and strength protocol 80% 1 RM) and body segments (elbow flexion [UL] and knee extension [LL]).
  RMSSD: root mean square of the successive differences between the RR intervals in the record, divided by the number of RR intervals in a given time minus one RR interval SDNN: standard deviation of all normal RR intervals.
Acute responses of the Autonomic Nervous System post Resistance Training of the geometric indices of Heart Rate Variability | the moments before and immediately after Resistance Training, performed with different intensities (endurance and strength) and body segments (UL and LL).
  Understand the effect of acute responses of the geometric indices of Heart Rate Variability, SD1, SD2, comparing the behavior of these indices of in rest periods and immediate recovery after effort. Besides, to analyze the changes observed when applying different training intensities (endurance protocol 40% 1RM, and strength protocol 80% 1 RM) and body segments (elbow flexion [UL] and knee extension [LL]).
  SD1: standard deviation of diagonal points SD2: standard deviation from longitudinal points
Acute responses of the Autonomic Nervous System post Resistance Training of the frequency domain of Heart Rate Variability, | the moments before and immediately after Resistance Training, performed with different intensities (endurance and strength) and body segments (UL and LL).
  Understand the effect of acute responses of the frequency domain of Heart Rate Variability, LF anf HF, both calculated in absolute (ms2) and normalized units (nu), comparing the behavior of these indices of in rest periods and immediate recovery after effort. Besides, to analyze the changes observed when applying different training intensities (endurance protocol 40% 1RM, and strength protocol 80% 1 RM) and body segments (elbow flexion [UL] and knee extension [LL]).
  LF: spectral components of low frequency, 0.04 - 0.15Hz HF: spectral components of high frequency, 0.15 - 0.40 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, Professor, Study Director — Universidade Estadual Paulista - FCT/UNESP
Locations (2):
- Brazil (2):
  - Luiz Carlos Marques Vanderlei, Presidente Prudente, São Paulo
  - Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo

REFERENCES:
- See also: Catai, A. M., Pastre, C. M., Godoy, M. F. de, Silva, E. da, Takahashi, A. C. de M., & Vanderlei, L. C. M. (2019). Heart rate variability: are you using it properly? Standardisation checklist of procedures. Brazilian Journal of Physical Therapy — http://pubmed.ncbi.nlm.nih.gov/30852243/
- See also: Collins H., Booth J.N., Duncan A., Fawkner S., Niven A. The effect of resistance training interventions on 'The Self' in Youth: a systematic review and meta-analysis. — http://sportsmedicine-open.springeropen.com/articles/10.1186/s40798-019-0205-0
- See also: Evans JW. Periodized resistance training for enhancing skeletal muscle hypertrophy and strength: a mini review. — http://www.frontiersin.org/articles/10.3389/fphys.2019.00013/full
- See also: Kingsley, J. D., & Figueroa, A. (2016). Acute and training effects of resistance exercise on heart rate variability. — http://pubmed.ncbi.nlm.nih.gov/25524332/
- See also: Guedes DP, Lopes CC, Guedes JERP. (2005). Reprodutibilidade e validade do Questionário Internacional de Atividade Física em adolescentes. — https://www.scielo.br/scielo.php?script=sci_arttext&pid=S1517-86922005000200011
- See also: Vanderlei, Luiz Carlos Marques, Pastre, C. M., Hoshi, A., Dias, T., & Fernandes, M. (2009). Noções básicas de variabilidade da frequência cardíaca e sua aplicabilidade clínica. — https://www.scielo.br/scielo.php?script=sci_arttext&pid=S0102-76382009000200018
- See also: American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009;41(3):687-708. doi:10.1249/MSS.0b013e3181915670 — https://pubmed.ncbi.nlm.nih.gov/19204579/